CLINICAL TRIAL: NCT07122726
Title: Additional Effects of Proprioceptive Neuromuscular Facilitation With Otago Exercises on Fall Risk in Diabetes Mellitus Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/83
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Postural Balance; Fall Risk; Diabetes (DM); Fear of Falling; Sensory Function; Diabetic Neuropathy Peripheral; Proprioceptive Neuromuscular Facilitation
Keywords: Balance; Fall risk; Fear of fall; sensory function; Otago Exercises; Proprioceptive neuromuscular facilitation; Diabetic Peripheral Neuropathy; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Otago with PNF (Experimental): Otago exercise plan is comprised set of 14 exercises including strengthening and balance exercises. The strengthening exercises include strengthening of Knee Flexors, Knee Extensors, Hip-abductors Ankle dorsiflexors and ankle planter flexors and the balance exercises include following activities: Knee Bends Backward Walking, Walking and Turning Around, Sideways Walking, Tandem Stance, Tandem Walk, One Leg stance, Heel Walking, Toe Walking, Heel toe walk backwards, Sit to stand, Stair Walking The PNF pattern includes includes incorporating diagonal patterns, reversal of agonists, and combination of isotonic to enhance neuromuscular control. These techniques will be applied progressively based on patient response and capability. The gradually increasing resistance throughout the range of motion will be applied. The exercise intervention consists of 6 levels.
  These exercises will be performed for a duration 6 weeks and will be performed thrice for a period of 40/50 minutes.
  Interventions: Procedure: Otago and PNF exercise
- Otago Exercise (Active Comparator): Otago exercise plan is comprised set of 14 exercises including strengthening and balance exercises. The strengthening exercises include strengthening of Knee Flexors, Knee Extensors, Hip-abductors Ankle dorsiflexors and ankle planter flexors and the balance exercises include following activities: Knee Bends Backward Walking, Walking and Turning Around, Sideways Walking, Tandem Stance, Tandem Walk, One Leg stance, Heel Walking, Toe Walking, Heel toe walk backwards, Sit to stand, Stair Walking These exercises will be performed for a duration 6 weeks and will be performed thrice for a period of 40/50 minutes.
  Interventions: Procedure: Otago Exercise

INTERVENTIONS:
Procedure: Otago and PNF exercise — Otago Exercise:
  This 6-week protocol focuses on strengthening and balance exercises. It starts with supported exercises and progresses to unsupported ones. Exercises include knee flexors, extensors, and hip abductors with ankle weights, ankle plantar and dorsiflexors, knee bends, backward stepping, walking and turning, sideways walking, tandem stance, and one-leg stance. Repetitions increase over time, from 10-20 reps with support to 30 reps without support.
  PNF Exercise The PNF protocol consists of 6 levels, progressing from simple to complex exercises. Level 1 involves D1/D2 patterns for ankle and hip with light resistance, while Level 2 focuses on seated D1/D2 patterns for the lower limb. Levels 3-6 introduce more dynamic exercises, including arm reaches while standing, PNF walking, dynamic step-ups, walking on unequal terrain, and obstacle navigation. The protocol emphasizes approximation, stabilization, resistance, and dynamic reversals to improve proprioception & balance.
  Arms: Otago with PNF
Procedure: Otago Exercise — Knee Flexors, Knee Extensors, Hip-abductors- 10 reps of each Exercise with ankle weights to provide muscle resistance. For ankle planter flexors and dorsi flexors starting from 20 repetitions at week 1 with hold support and ending at 30 repetitions without any support on 6th week. For knee bends starting with 10 reps at week 1 and ending at 30 reps without support at 6th week. Backward stepping 10 times 2 steps backward at week 1 progressing to 10 times x 4 Steps x No Support at week 6 gradually. Walking and Turning Around- (make a figure of 8), twice, first with support and then without support. Sideways Walking- 10 steps, 4 times x first with support and then without support over the time of 6 weeks. Tandem Stance- 10 seconds first with support and then without support. Tandem Walk/ 20 reps first with support and then without support over the period of 6 weeks.
  Arms: Otago Exercise

SUMMARY:
Diabetes Mellitus is considered as one of the most prevalent issues among global population and 50% of all the diabetic patients particularly diabetes type II develop peripheral neuropathy. Diabetic Peripheral Neuropathy (DPN) affects feet and legs first, followed by the hands and arms.

This study will involve two groups, one performing the Otago Exercise Program, and the other performing a combined PNF and Otago exercise protocol. This study aims to assess the additional effects of Proprioceptive Neuromuscular Facilitation with Otago Exercise Program on Risk of fall which will be assessed by assessing balance, Fear of Fall and Sensory Function.

Key outcome measures, including the Berg Balance Scale, Fall Efficacy Scale, Functional Reach test and Semmes Weinstein Monofilament Test will be used in evaluating the effectiveness of the exercise interventions. The participants would be screened through Michigan Neuropathy Screening Instrument and Berg Balance scale for inclusion criteria, and outcome measures will be assessed by using Berg Balance Scale, Fall efficacy scale, Functional Reach Test and Semmes Weinstein Monofilament testing method on the day of starting the intervention and on the last day of intervention. Intervention will be given for a total of 40-50 minutes per session, 3 sessions/week for consecutive 6 weeks And than the data will be recorded at the end of 6 weeks again.

DETAILED DESCRIPTION:
The occurrence of diabetes mellitus (DM) is continually rising and has become one of the most evidently emerging chronic disease globally. One of the major consequence of Diabetes Mellitus is Diabetic Peripheral Neuropathy (DPN) which is associated with symptoms like pain, tingling, numbness, paresthesia, balance problems and falls etc. The overall pooled prevalence of diabetic peripheral neuropathy in Pakistan was estimated to be 43.16%. Diabetic Peripheral Neuropathy (DPN) causes weakness, numbness and pain in the hands and feet. Sensory disturbance leads to loss of vibration, pressure, temperature and pain. In addition people with DPN experience muscle weakness, loss of ankle reflexes, drop balance, loss of coordination etc.

Proprioceptive Neuromuscular Facilitation (PNF) is a system that uses diagonal and spiral movements, and different techniques like Reversal of Antagonists, Dynamic Reversals, and Rhythmic Initiation intended at facilitating, strengthening, gaining control of movement. The Otago Exercise Program was originally designed to prevent falls by improving balance. It involves leg muscle strengthening, walking and balance retraining exercises designed specifically to prevent falls and improve balance.

This study offers a novel approach by comparing the effects of the Otago Exercise Program with a combined PNF and Otago exercise protocol, targeting multiple domains crucial for functional improvement in DPN patients. This study is a randomized control trial and will be conducted for a duration of year, and Non-probability Convenient Sampling technique will be used for the study. The exercises will be performed for 6 weeks and thrice a week for 40-50 minutes on sample of 30 selected through G Power.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type 2 patients
* 50-75 years of age
* Both Males and Female Gender
* Duration of diabetes more than 5 years
* Participants positive for Michigan Neuropathy Screening Instrument
* Patients having berg balance scale score >20

Exclusion Criteria:

* Surgical procedure involving knee, ankle, or hip joints.
* Foot Ulcers and Deformities.
* Diagnosis of neurological diseases (CVA, MS, Parkinson disease etc.) besides DPN.
* Absence of Visual Impairment and Hearing loss Patients having comprehension difficulties
* Physical disability that prevents from performing the exercises

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Balance | 6 weeks
  Balance will be assessed using berg balance scale. total score is 58. low fall risk is 0-20, moderate risk 20-40, High risk 41-58
Fear of fall | 6 weeks
  The Falls Efficacy Scale-International (FES-I) will be used to measures the level of concern about falling. The level of concern is measured on a four point Likert scale (1=not at all concerned to 4=very concerned).
Balance | 6 weeks
  The functional reach test will be performed to analyze dynamic balance. The patients will be instructed to position themselves with their body perpendicular to the wall but not touching the wall, with shoulders flexed at 90°, elbows extended, and hands closed. The assessor will record the starting position at the 3rd metacarpal head on the yardstick and then instruct the patient to reach as far as they can without taking a step, and the distance will be measured between the initial measurements to the final measurement.
Sensory function | 6 weeks
  The SEMMES WEINSTEIN MONOFILAMNET TESTING is considered a simple and inexpensive touch threshold test and is widely used by clinicians to evaluate sensory disturbances of neuropathic diseases. With the patient's eyes closed, monofilament is applied perpendicularly in a steady manner until the filament bends. Use a smooth motion to touch the skin with the filament, bend the filament for a full second, than lift from the skin. Patient raises hand to indicate that the monofilament touch sensation is perceived.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan